CLINICAL TRIAL: NCT01484184
Title: Tri-therapy (SPINALON)-Elicited Spinal Locomotor Network Activation: Phase I-IIa Clinical Trial in Patients With Chronic Spinal Cord Injury
Brief Title: Study to Assess Safety, Tolerability and MTD of a Central Pattern Generator-activating Tritherapy (SPINALON) in Patients With Chronic Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nordic Life Science Pipeline Inc. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: SPIN-01
Record Dates: First submitted 2011-11-25; First posted 2011-12-02 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Spinal Cord Injury
Keywords: Completely paralyzed; Chronically injured; Central Pattern Generator; Locomotion; Secondary complications; Activity-based training; Treadmill training; Spinal cord injury; Paraplegia; Tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia | interventions — Buspirone; Levodopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- buspirone or levodopa/carbidopa (Active Comparator): Another 2-arm design will be tested composed of 16 subjects receiving drug A or drug B at MTD dose of the combined study drug as identified in the previous 2-arm groups.
  Interventions: Drug: SPINALON (buspirone + levodopa + cardidopa)
- Placebo (Placebo Comparator): First, a 2-arm design will be used, the first arm being composed of 3 subjects receiving the lowest dose of SPINALON, the second arm being composed of 1 subject receiving a placebo. This 2-arm design will be repeated consecutively with increasing doses, as long as the dose is well tolerated. Six (6) groups are expected to be tested with this 2-arm design.
  Interventions: Drug: SPINALON (buspirone + levodopa + cardidopa)

INTERVENTIONS:
Drug: SPINALON (buspirone + levodopa + cardidopa) — The proposed study is a combination of 1 and 2-arm designs. First, a 2-arm design will be used, the first arm being composed of 3 subjects receiving the lowest dose of the study drug, and the second arm being composed of 1 subject receiving a placebo. This 2-arm design will be repeated consecutively (not simultaneously) with increasing doses of SPINALON, as long as the dose is well tolerated. Six (6) groups are expected to be tested with this 2-arm design.This will be followed by a 2-arm composed of 1 group with 1 subject receiving placebo and 1 larger group (10 subjects) who will receive SPINALON at MTD as identified in the previous 2-arm groups.
  Other Names: Apo-Buspirone 10 mg tablets (DIN 02211076); Sinemet 100/25 mg tablets (DIN 00513997)

SUMMARY:
As a first-in-class (Central Pattern Generator or CPG activator) approach, this tritherapy candidate called SPINALON has been identified and is currently under development for its capacity to temporarily induce episodes of involuntary locomotor movements. The primary objective of this Phase I/IIa study is to assess safety and tolerability of a single escalating dose of SPINALON (levodopa + carbidopa + buspirone) in chronic spinal cord-injured patients. As a secondary objective, preliminary evidence of efficacy will also be sought.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is generally considered as an irreversible condition for which no curative treatment has yet been found. A recent study sponsored by the Christopher & Dana Reeve Foundation revealed an incidence ranging between 40 and 60 cases per million population and a prevalence estimated to be several times greater (new data: 1,275,000 cases) than previously reported(previous data: 200,000 cases).

SPINALON (levodopa + carbidopa + buspirone) was discovered by Dr. Guertin and colleagues as a drug treatment candidate that can acutely elicit temporarily (lasting approximately 30-60 minutes) episodes of CPG activity and corresponding powerful weight-bearing hindlimb stepping in completely SCI subjects (preclinical efficacy data obtained from mice and turtles completely spinal cord transected thoracically).

As such, SPINALON is currently being developed to become a chronic treatment (physical activity-based approach driven pharmacologically) against the multiple health problems or so-called 'secondary complications' associated specifically with the lack of physical activity (sarcopenia, osteoporosis, cardiovascular problems, dyslipidemia, obesity, type II diabetes, anemia, immune system deficiency, deep vein cloth, depression, etc.).

This study is a randomized, placebo-controlled, double-blind, single dose escalation study with fifty-one (51) patients who will receive either placebo capsules(starch) or capsules with buspirone only, levodopa/carbidopa only or buspirone/levodopa/carbidopa (SPINALON).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of complete or motor-complete SCI (ASIA-A, ASIA-B)
* Chronically injured (at least 3 months post-injury)
* Paraplegic (within T1-T12) or tetraplegic (within C3-C8)
* In relatively good health condition (no significant bed sore, urinary tract infection)
* 18-65 years of age
* Men and women
* Quebec Province residents only

Exclusion Criteria:

* With unclear diagnosis
* Displayed a form of involuntary rhythmic leg muscle activity (restless leg syndrome, spontaneous activity in supine position, etc.) in the last 3 months prior to this study.
* Acute or subacute stage (within 1 day and 3 months post-injury)
* Non-traumatic (e.g., multiple sclerosis, syringomyelia, spinal tumor,etc.)
* Are given monoamine oxidase (MAO) inhibitors (two weeks prior and after Spinalon administration)
* Had seizures
* Had tumor(s) (malignant or non-malignant) or in situ carcinoma in the last five (5) years
* Allergic or hypersensitive to buspirone, levodopa or carbidopa
* Can not take sympathomimetic amines (e.g., epinephrine, pseudoephedrine)
* Currently suffering of heart problems, blood related diseases, endocrine disease, liver disease, lung disease, or kidney disease
* Receiving antihypertensive drugs
* Receiving tricyclic antidepressant
* Receiving dopamine D2 receptor antagonists (e.g., phenothiazines, butyrophenones, risperidone)
* Receiving phenytoin and papaverine
* With glaucoma
* With psychiatric or mental disorder(s)
* Had gastrointestinal ulcer(s) in the last five (5) years
* Pregnant or lactating woman (all women between 18 and 50 year-old not yet confirmed as pregnant, will be tested (urine test - TestPak Plus, Abbott Laboratories) on medical exam-day due to the teratogenic potential of levodopa/carbidopa.
* Children (younger than 18 year-old) or elderly (older than 65 year-old)
* Not resident of Quebec Province

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Heart rate | Steadily during 4 hours post-single administration vs pre-administration
  Heart rate as a safety measure will be measured as beats per minute during 4 hours post-administration during the only administration
Tolerability of common AEs | During 4 hours post-single administration vs pre-administration
  Frequent AEs such as nausea and hypotension will be specifically measured to assess tolerability and maximum tolerated dose. No more than 20% of subjects experiencing nausea with > grade 2 severity. Dose schedule without ≥ grade 3 hypotension. No potentiation of other AEs possibly found for each molecule administered separately
Pharmacokinetics | 15, 30, 60, 120 and 240 min post-administration vs pre-administration
  Blood samples will be repeatedly obtained post-administration on the day of testing. HPLC analysis will be conducted to assess typical PK values (Cmax, Tmax, AUC) in order to determine whether or not the known PK profile of each active molecule (levodopa, carbidopa, buspirone) is changed once administered concomitantly (SPINALON)
Blood pressure | During 4 hours post-single administration vs pre-administration
  Systolic and diastolic blood pressure values as a safety measure will be measured as mmHg during 4 hours
Respiration rate | During 4 hours post-single administration vs pre-administration
  Respiration rate as number per minute will be measured as a safety issue during 4 hours post-administration compared with baseline value pre-administration on the day of testing
Oxygen saturation | During 4 hours post-single administration vs. pre-administration
  Oxygen saturation measured as CO2 level and O2 level in percentage will be measured on the day of testing during 4 hours post-administration compared with baseline level (pre-administration)
Temperature | During 4 hours post-single administration vs. pre-administration
  Temperature measured in degrees Celsius will be measured during 4 hours post-administration on the day of testing compared with baseline value (pre-administration)
Change in hematology and biochemistry laboratory parameters | Once at 4 hours post-single administration vs pre-administration
  Blood samples at 4 hours post-administration will be analyzed for standard hematology (CBC) and biochemistry (liver and kidney markers) values and compared with baseline values (medical exam day sample).

SECONDARY OUTCOMES:
Occurrence of rhythmic leg EMGs | During 2 hours post-administration vs pre-administration
  EMG activities of leg muscles will be measured with surface electrodes during 2 hours post-administration on the day of testing compared with baseline values pre-administration. Possible occurrence of involuntary rhythmic and bilateral movements assessed quantitatively will be sought.

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Radhakrishna, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Pierre Guertin, Ph.D., Study Director — Nordic Life Science Pipeline/Université Laval
Locations (1):
- McGill University Health Centre (Montreal General Hospital), Montreal, Quebec, Canada

REFERENCES:
- [Background] Guertin PA, Ung RV, Rouleau P, Steuer I. Effects on locomotion, muscle, bone, and blood induced by a combination therapy eliciting weight-bearing stepping in nonassisted spinal cord-transected mice. Neurorehabil Neural Repair. 2011 Mar-Apr;25(3):234-42. doi: 10.1177/1545968310378753. Epub 2010 Oct 15. PMID 20952632
- [Background] Guertin PA, Ung RV, Rouleau P. Oral administration of a tri-therapy for central pattern generator activation in paraplegic mice: proof-of-concept of efficacy. Biotechnol J. 2010 Apr;5(4):421-6. doi: 10.1002/biot.200900278. PMID 20349462
- [Background] Guertin PA. The mammalian central pattern generator for locomotion. Brain Res Rev. 2009 Dec 11;62(1):45-56. doi: 10.1016/j.brainresrev.2009.08.002. Epub 2009 Aug 29. PMID 19720083
- [Background] Lapointe NP, Rouleau P, Ung RV, Guertin PA. Specific role of dopamine D1 receptors in spinal network activation and rhythmic movement induction in vertebrates. J Physiol. 2009 Apr 1;587(Pt 7):1499-511. doi: 10.1113/jphysiol.2008.166314. Epub 2009 Feb 9. PMID 19204052
- [Background] Lapointe NP, Guertin PA. Synergistic effects of D1/5 and 5-HT1A/7 receptor agonists on locomotor movement induction in complete spinal cord-transected mice. J Neurophysiol. 2008 Jul;100(1):160-8. doi: 10.1152/jn.90339.2008. Epub 2008 May 14. PMID 18480366
- [Background] Landry ES, Lapointe NP, Rouillard C, Levesque D, Hedlund PB, Guertin PA. Contribution of spinal 5-HT1A and 5-HT7 receptors to locomotor-like movement induced by 8-OH-DPAT in spinal cord-transected mice. Eur J Neurosci. 2006 Jul;24(2):535-46. doi: 10.1111/j.1460-9568.2006.04917.x. Epub 2006 Jul 12. PMID 16836640